CLINICAL TRIAL: NCT02245399
Title: Canola Enriched Mediterranean Type Weight Loss Diet in Type 2 Diabetes
Brief Title: Canola-Mediterranean Diet Study in T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other); Laval University (Other); University of Manitoba (Other); Canola Council of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB# 14-086; CFC/Fund 200134/496744 (Other: Canola Council of Canada)
Record Dates: First submitted 2014-09-05; First posted 2014-09-19 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes; Obesity; Overweight; Cardiovascular Diseases
Keywords: Weight loss; Diabetes; Cardiovascular disease (CVD) risk; Weight loss diet; mediterranean type diet; Canola oil; Low-carbohydrate diet; Glycemic index
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight; Cardiovascular Diseases; Weight Loss; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A canola oil enriched mediterranean diet (Experimental): Participants will be advised to consume, a low-carbohydrate diet (26-32% of calories), high in vegetable protein (28-32%) and fat (41-45%) with canola as the major component (10%). Carbohydrate sources will feature viscous fiber-containing foods (including psyllium cereal, oats and barley) and low-starch vegetables (emphasizing okra and eggplant) for the relatively limited amount of carbohydrate.
  Interventions: Behavioral: A canola oil enriched mediterranean diet
- A high wheat fiber diet (Active Comparator): Participant will be advised to consume a high carbohydrate diet (58% carbohydrate, 16% protein and 25% fat) emphasizing whole wheat/whole grain cereals and increased high fiber alternatives, with fruits and vegetables.
  Interventions: Behavioral: A high wheat fiber diet

INTERVENTIONS:
Behavioral: A canola oil enriched mediterranean diet — The diet will be provided at 60% of calories estimated for stable body weight to encourage weight loss. A high protein canola oil-enriched test bread will be provided as a supplement.
  Other Names: A mediterranean weight-reducing diet emphasizing canola oil; Eco-Atkins diet; Low carbohydrate dietary portfolio
  Arms: A canola oil enriched mediterranean diet
Behavioral: A high wheat fiber diet — The diet will be provided at 60% of calories estimated for stable body weight to encourage weight loss. A whole wheat control bread will be provided as a supplement to participants
  Other Names: DASH-type diet
  Arms: A high wheat fiber diet

SUMMARY:
The purpose of the study is to assess whether a Mediterranean-type weight-loss diet, enriched with canola oil, high in plant protein, and low in carbohydrates will produce blood sugar control, reduce coronary heart disease (CHD) risk factors and maximize weight loss, better than conventional higher carbohydrate diets in overweight diabetic patients.

DETAILED DESCRIPTION:
The investigators plan to assess the effects of increasing both canola oil and plant protein foods while reducing carbohydrate intake in the context of a Mediterranean type diet on weight loss, glycemic control and cardiovascular risk factors in type 2 diabetes.

Obesity rates in Western nations have shown a dramatic rise in the last 20 years and diabetes rates have doubled, a trend which is predicted to be repeated over the next 20 years. In Canada the predicted cost to the healthcare system in only 7 years will rise to $17 billion. Weight loss diets (such as Atkins, Eddies, South Beach and Zone) emphasizing carbohydrate restriction have become increasingly popular for the prevention and treatment of diabetes. As a result, lower carbohydrate diets are being selected by health conscious members of the general population including those with diabetes. Because such diets in effect promote a high intake of protein from animal sources, even in the presence of weight loss, serum cholesterol levels rise due to increased cholesterol and saturated fat intake; and a further rise in serum lipids is likely to occur in the long term when weight loss has ceased. On the other hand, lower carbohydrate dietary patterns that are higher in plant rather than animal fat and proteins have been associated with improved blood lipids and reduced risk of heart disease and type 2 diabetes.

The investigators have therefore planned a study in which a weight reducing low carbohydrate, Mediterranean type diet that is high in plant proteins and canola oil will be compared to a weight reducing high cereal fibre diet in a 3 month study. 150 overweight and obese participants with type 2 diabetes will be randomized to one of 2 treatments.

Study visits will be as follows: weeks -2, 0 (for randomization), 2, 4, 8, 10 and 12. Body measurements, blood pressure and blood samples will be taken at each visit except week 2. The week 2 visit will be mainly for reinforcement of dietary advice; also body weight will be measured and blood drawn for fast glucose and HbA1c. Diet records will be reviewed at all visits. 24 hour urine samples will be collected at week 0 and week 12.

On completion of the 12 week study, participants will be given the option of continuing on the same diet or trying the opposite diet for a further 12 weeks. Visits will be every 4 weeks for a total of 3 visit. Body measurements, blood pressure and blood samples will be taken during these visits as in the initial 12 week study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with type 2 diabetes diagnosed for more than 6 months
* BMI >27 (non-Asians); BMI >25 (Asians)
* HbA1c between 6.5% and 8.5% at screening, and at the preparation visit before starting diet
* on a stable prescribed dose of oral diabetes medication for at least 2 months
* on a stable dose of lipid medication for at least 2 weeks, if prescribed
* on a stable dose of blood pressure medication for at least 1 week, if prescribed
* have a family physician
* can keep written food records, with the use of a digital scale

Exclusion Criteria:

Individuals with the following characteristics/conditions will be excluded

* on insulin
* on steroids
* on warfarin (Coumadin)
* GI disease (gastroparesis, celiac, colitis, Crohn's disease, Inflammatory Bowel Syndrome)
* history of cancer, except non-melanoma skin cancer (basal cell, squamous cell)
* major cardiovascular event (stroke, myocardial infarction) in past 6 months
* major surgery in past 6 months
* major debilitating disorder
* liver disease (AST or ALT> 3x the upper limit of normal) except non-alcoholic fatty liver (NAFL) disease or non-alcoholic steatohepatitis (NASH).
* hepatitis B or C
* renal failure (creatinine > 150 mmol/L)
* serum triglycerides >4.5mmol/L
* acute or chronic infections (bacterial or viral)
* chronic inflammatory diseases (e.g. lupus, ulcerative colitis)
* blood pressure >145/90, unless approved by their family physician
* alcohol consumption >2 drinks/d
* food allergies to wheat, canola, or other study food components
* any condition determined by the investigators to make the subject unsuitable for the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
change in HbA1c | Measured at weeks -2, 0, and then at weeks 8, 10 and 12
  The baseline HbA1c will be the average HbA1c of weeks -2 and week 0. The end HbA1c will be the average HbA1c of weeks 8, 10 and 12. Change will be the difference between the end and baseline values

SECONDARY OUTCOMES:
Change in body weight | baseline (week 0) and end (week 12)
blood glucose | At weeks 0, 2, 4, 8, 10 and 12
Serum lipids: total cholesterol, LDL-chol, HDL-chol and Triglycerides | At weeks 0, 4, 8, 10 and 12
Blood pressure | At weeks 0, 4, 8, 10 and 12
24-hour Ambulatory blood pressure profile | At weeks -1 and 12
  Measurement will be done using a non-invasive SpaceLabs 90217 Ambulatory BP monitor
diet history | At weeks 0, 2, 4, 8, 10 and 12
  7-day food records brought in at weeks 0, 2, 4, 8, 10 and 12 will be analyzed for macro and micro nutrient intakes.
C-reactive protein | At weeks 0 and 12
Cholesterol absorption | At weeks -1 and 12
  This is an optional sub-study that will be carried out prior to the first and last weeks of the 12 week study. On day 1 (a Monday) of the week -1 and last weeks of the study after an overnight 12hr fast, blood will be drawn and participants will be asked to ingest 75mg of the stable carbon isotope [3, 4-13C] cholesterol dissolved in 5g of margarine and spread on half of an English muffin. Subsequent blood draws will be taken after an overnight 12hr fast, at 48 h (a Wednesday) and 72 h (a Thursday) after ingestion of the labeled cholesterol.
change in LDL particle size | Weeks 0 and 12
  LDL particle size at weeks 0 and 12 will be determined by assessing their electrophoretic characteristics obtained by non-denaturing polyacrylamide gradient (2-16%) gel electrophoresis of serum
urinary analyses | week 0 and week 12
  24 hr urine samples will be analyzed for creatinine, urea, C-peptide, minerals, electrolytes and other dietary biomarkers

OTHER OUTCOMES:
Satiety | at weeks 0, 2, 4, 8, 10 and 12
  Using a 9-point bipolar semantic scale where -4 is extremely hungry, 0 is neutral and +4 is uncomfortably full, participants will rate their overall feeling of satiety for the previous week.
Taste (palatability) of the study diets, breads and other supplements given | At weeks 2, 4, 8, 10 and 12
  Using a scale of 1 (strongly dislike) to 10 (like very much), participants will rate the taste (palatability) of the study diet and supplements including study breads, vegan 'meats' and egg products.
The Medical Outcomes Study 36-Item Short Form Questionnaire (SF-36) | At weeks 0 and 12
  Survey on quality of life
Genetic whole genome testing | Week 0 or any other time point
  One time sample collection of buffy coat (from white cells) for future study on gene, diet and chronic disease relationship.
complete blood count (CBC) | Week 0 and week 12
  Health check at start and end of study
Renal function test | week 0 and week 12
  Health check at start and end of study
Liver function test | week 0 and week 12
  Health check at start and end of study
Prostatic specific antigen (PSA) | week 0 and week 12
  Male participants will undergo this test.
sustainability of diet | week 10 and week 12
  using a scale of 1 (study diet will be very difficult to sustain) to 10 (study diet will be very easy to sustain) participants will assess how sustainable their assigned diet will be on a long-term basis.
Testosterone level | week 0 and week 12
  Male participants will undergo this test
Estradiol level | week 0 and week 12
  Female participants will undergo this test

CONTACTS AND LOCATIONS:
Overall Officials: David J Jenkins, MD, Principal Investigator — St. Michael's Hospital / University of Toronto; Cyril Kendall, PhD, Study Director — University of Toronto; Vladimir Vuksan, PhD, Study Director — Unity Health Toronto; Peter Jones, PhD, Study Director — University of Manitoba; Benoit Lamarche, PhD, Study Director — Laval University
Locations (3):
- Canada (3):
  - Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba
  - Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario
  - Institute of Nutraceuticals and Functional Foods, Laval University, Québec, Quebec

REFERENCES:
- [Background] Alhassan S, Kim S, Bersamin A, King AC, Gardner CD. Dietary adherence and weight loss success among overweight women: results from the A TO Z weight loss study. Int J Obes (Lond). 2008 Jun;32(6):985-91. doi: 10.1038/ijo.2008.8. Epub 2008 Feb 12. PMID 18268511
- [Background] Anderson JW, Randles KM, Kendall CW, Jenkins DJ. Carbohydrate and fiber recommendations for individuals with diabetes: a quantitative assessment and meta-analysis of the evidence. J Am Coll Nutr. 2004 Feb;23(1):5-17. doi: 10.1080/07315724.2004.10719338. PMID 14963049
- [Background] Shai I, Schwarzfuchs D, Henkin Y, Shahar DR, Witkow S, Greenberg I, Golan R, Fraser D, Bolotin A, Vardi H, Tangi-Rozental O, Zuk-Ramot R, Sarusi B, Brickner D, Schwartz Z, Sheiner E, Marko R, Katorza E, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; Dietary Intervention Randomized Controlled Trial (DIRECT) Group. Weight loss with a low-carbohydrate, Mediterranean, or low-fat diet. N Engl J Med. 2008 Jul 17;359(3):229-41. doi: 10.1056/NEJMoa0708681. PMID 18635428
- [Background] Jenkins DJ, Wong JM, Kendall CW, Esfahani A, Ng VW, Leong TC, Faulkner DA, Vidgen E, Greaves KA, Paul G, Singer W. The effect of a plant-based low-carbohydrate ("Eco-Atkins") diet on body weight and blood lipid concentrations in hyperlipidemic subjects. Arch Intern Med. 2009 Jun 8;169(11):1046-54. doi: 10.1001/archinternmed.2009.115. PMID 19506174
- [Background] Guariguata L, Whiting D, Weil C, Unwin N. The International Diabetes Federation diabetes atlas methodology for estimating global and national prevalence of diabetes in adults. Diabetes Res Clin Pract. 2011 Dec;94(3):322-32. doi: 10.1016/j.diabres.2011.10.040. Epub 2011 Nov 17. PMID 22100977
- [Background] Kris-Etherton P, Eckel RH, Howard BV, St Jeor S, Bazzarre TL; Nutrition Committee Population Science Committee and Clinical Science Committee of the American Heart Association. AHA Science Advisory: Lyon Diet Heart Study. Benefits of a Mediterranean-style, National Cholesterol Education Program/American Heart Association Step I Dietary Pattern on Cardiovascular Disease. Circulation. 2001 Apr 3;103(13):1823-5. doi: 10.1161/01.cir.103.13.1823. No abstract available. PMID 11282918
- [Background] Sacks FM, Bray GA, Carey VJ, Smith SR, Ryan DH, Anton SD, McManus K, Champagne CM, Bishop LM, Laranjo N, Leboff MS, Rood JC, de Jonge L, Greenway FL, Loria CM, Obarzanek E, Williamson DA. Comparison of weight-loss diets with different compositions of fat, protein, and carbohydrates. N Engl J Med. 2009 Feb 26;360(9):859-73. doi: 10.1056/NEJMoa0804748. PMID 19246357
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Jenkins DJ, Wong JM, Kendall CW, Esfahani A, Ng VW, Leong TC, Faulkner DA, Vidgen E, Paul G, Mukherjea R, Krul ES, Singer W. Effect of a 6-month vegan low-carbohydrate ('Eco-Atkins') diet on cardiovascular risk factors and body weight in hyperlipidaemic adults: a randomised controlled trial. BMJ Open. 2014 Feb 5;4(2):e003505. doi: 10.1136/bmjopen-2013-003505. PMID 24500611
- [Background] Gremaud G, Piguet C, Baumgartner M, Pouteau E, Decarli B, Berger A, Fay LB. Simultaneous assessment of cholesterol absorption and synthesis in humans using on-line gas chromatography/ combustion and gas chromatography/pyrolysis/isotope-ratio mass spectrometry. Rapid Commun Mass Spectrom. 2001;15(14):1207-13. doi: 10.1002/rcm.365. PMID 11445904
- [Derived] Jenkins DJ, Jones PJ, Abdullah MM, Lamarche B, Faulkner D, Patel D, Sahye-Pudaruth S, Paquette M, Bashyam B, Pichika SC, Kavanagh ME, Patel P, Liang F, Brown R, Zhao T, Phan M, Mathiyalagan G, Tandon S, Vuksan V, Jovanovski E, Sievenpiper JL, Kendall CW, Leiter LA, Josse RG. Low-carbohydrate vegan diets in diabetes for weight loss and sustainability: a randomized controlled trial. Am J Clin Nutr. 2022 Nov;116(5):1240-1250. doi: 10.1093/ajcn/nqac203. Epub 2023 Feb 10. PMID 36156115